CLINICAL TRIAL: NCT00477724
Title: Incidence of Latent Pulmonary Hypertension in Patients With Chronic Thromboembolic Pulmonary Hypertension After Endarterectomy and Influence of Exercise and Respiratory Therapy
Brief Title: Latent Pulmonary Hypertension (PH) in Chronic Thromboembolic Pulmonary Hypertension (CTEPH )After Endarterectomy and Influence of Exercise and Respiratory Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REHA/CTEPH
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension; Chronic Thromboembolic Pulmonary Hypertension
Keywords: latent
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Exercise; Respiratory Therapy

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- sedentary control group (Placebo Comparator): patients are treated by conventional rehabilitation
  Interventions: Other: sedentary control group
- exercise and respiratory therapy (Active Comparator): rehabilitation with exercise and respiratory therapy
  Interventions: Behavioral: exercise and respiratory therapy

INTERVENTIONS:
Behavioral: exercise and respiratory therapy — exercise and respiratory therapy for three weeks in-hospital and 15 weeks at home
  Arms: exercise and respiratory therapy
Other: sedentary control group — control group with no specific training
  Arms: sedentary control group

SUMMARY:
Severe CTEPH leads to an impaired physical capacity and a restricted quality of life and poor prognosis.

Pulmonary endarterectomy represents the best choice as therapy, when the thrombi are located in the central pulmonary vessels and therefore can be operated. By this operation the pulmonary artery pressure can be normalised and the patients' survival improved. Up to now, after successful endarterectomy patients only receive anticoagulation.

Despite operation many patients remain symptomatic and are restricted in their physical capacity. Therefore a hypothesis of this project is that most of the patients, even after successful operation, show peripheral vascular remodelling with a ventilation-perfusion mismatch and elevated pulmonary pressure during exercise.

In this study we aim to analyse how many patients with CTEPH after endarterectomy show elevated pulmonary artery pressures at rest or during exercise and are limited in their physical capacity, hemodynamics, oxygen uptake and quality of life and need further therapy.

Another aim is to examine whether exercise and respiratory therapy may improve the patients postoperatively.

Therefore 30 patients with CTEPH > six months after endarterectomy, with ongoing restricted exercise capacity shall be included. After baseline examination in the University hospital Heidelberg the patients receive exercise and respiratory therapy for three weeks. The patients will receive further examinations at the end of rehabilitation after 3 weeks and after 15 weeks. All examinations include medical history, family history, physical examination, ECG and echocardiography at rest and during exercise, cardiopulmonary exercise testing, assessment of the respiratory muscle strength, the SF-36 questionnaire for quality of life, laboratory testing and MRI.

Rehabilitation will be conducted in the clinic for rehabilitation Koenigstuhl, Heidelberg. Participants will be randomised into two groups, a control group receiving a conventional therapy for three weeks, in which physical exertion is to be avoided and a training group with additional exercise and respiratory therapy.

ELIGIBILITY:
Inclusion Criteria:

* A Screening

  1. Informed consent
  2. Men and women 18 - 75 years
  3. Patients ≥ 6 months after endarterectomy because of chronic thromboembolic pulmonary hypertension (CTEPH)
* B Training

See A + all patients who showed a restricted physical capacity in the screening:

* Latent pulmonary hypertension
* Restricted physical capacity

Exclusion Criteria:

1. Pregnancy or lactation
2. Change in medication during the last 2 months
3. Patients with signs of right heart decompensation
4. Disease which affects the gait
5. Unclear diagnosis
6. Acute illness, infection, fever
7. Severe lung diseases with FEV1 <50% and TLC< 70% of reference

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2007-06; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in 6-Minute walking test | after 3 and 15 weeks compared to baseline
Change in quality of life | baseline and 15 weeks

SECONDARY OUTCOMES:
physical capacity in the ergometer test | baseline, 3 and 15 weeks
change of lung function during 6-minute walking test | baseline, 3 and 15 weeks
noninvasive hemodynamic parameters | baseline, 3 and 15 weeks
change of systolic pulmonary arterial pressure at rest and during exercise | baseline, 3 and 15 weeks
change of WHO functional class | baseline, 3 and 15 weeks
change of perfusion parameters (MRI) | baseline, 3 and 15 weeks
change of respiratory muscle function | baseline and 15 weeks
change of NTproBNP | baseline, 3 and 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Gruenig, MD, Principal Investigator — Thoraxclinic at the University Hospital Heidelberg
Locations (1):
- Thoraxclinic at the University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Mereles D, Ewert R, Lodziewski S, Borst MM, Benz A, Olschewski H, Grunig E. Effect of inhaled iloprost during off-medication time in patients with pulmonary arterial hypertension. Respiration. 2007;74(5):498-502. doi: 10.1159/000101953. Epub 2007 Apr 20. PMID 17449958